CLINICAL TRIAL: NCT06085872
Title: Testing the REThinkACADEMY Interventions in Prevention of Emotional Disorders in First Year College Students.
Brief Title: Testing the REThinkACADEMY Interventions in Prevention of Emotional Disorders in College Students.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Collaborators: The Executive Agency for Higher Education, Research, Development and Innovation Funding (Other)
Responsible Party: Principal Investigator, Oana David, Professor Ph.D of Clinical Psychology, Babes-Bolyai University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: REThink Academy- SMARTrial
Record Dates: First submitted 2023-10-03; First posted 2023-10-17 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-10

CONDITIONS: Emotion Regulation; Stress
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- PsyPills - Experimental (Experimental): Each recruited student randomized in the experimental group will receive the PsyPills app.
  Interventions: Behavioral: PsyPills
- MoodWheel - Monitoring (Active Comparator): The students randomized in the control group will complete the MoodWheel app.
  Interventions: Behavioral: MoodWheel
- REThink Life Game (Experimental): Students from experimental group who do not respond to PsyPills alone will play the REThink Life Game
  Interventions: Behavioral: REThink Life Game; Behavioral: PsyPills

INTERVENTIONS:
Behavioral: REThink Life Game — REThink Life Game is the therapeutic game that uses psychological science to help youths find their superhero emotional strengths! It is composed of four levels, each training a specific emotion regulation ability: emotion recognition, mindfulness and relaxation, cognitive change and positive bias.
  Arms: REThink Life Game
Behavioral: PsyPills — PsyPills is a self-help psycho-educational instrument intended to build stress resilience and to target (only) mild and transient negative mood states, alone or in combination with other methods/instruments.
  Psychological Pills (PsyPills) are inspired by Rational-Emotive & Cognitive-Behavioral Therapy (CBT/REBT), which has strong evidence for its efficacy/effectiveness in human development/health promotion and in the treatment of a variety of psychological conditions.
  The PsyPills app was tested in a pilot study and showed positive effects on reducing distress. The efficacy of the app adjunct to other therapeutic tools within the platform in our projects will be tested.
  Arms: PsyPills - Experimental; REThink Life Game
Behavioral: MoodWheel — Mood Wheel is a web and mobile-based app that uses experience sampling procedures for the assessment of current/previous distress and positive emotions. The aim of the app is to inquire about the valence, control and functionality of users' emotions.
  Arms: MoodWheel - Monitoring

SUMMARY:
Entry in the REThinkACADEMY trial will be based on the high distress range on a psychological validate instrument to assess stress. After participants are enrolled in the REThinkACADEMY trial and randomized, those in the experimental condition ill access a ecological momentary intervention (EMI) app for the prevention of emotional disorders for 4 weeks. In the second stage, for the non-responders to the ecological supportive intervention, the online game will be implemented while the rest of the groups will be monitored for another 4 weeks. At the next step, post-test outcomes assessment will be implemented. Long term assessments will be conducted at 6 months for the college student's naturalistic follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

* to a first year student enorlled in Babes-Bolyai University of Cluj-Napoca
* internet and PC access to complete the scales and game
* high level of distress based on PDa scores

Exclusion Criteria:

* no internet or PC access

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2024-12-25 (Actual)

PRIMARY OUTCOMES:
Emotion regulation | baseline, pre-intervention
  Emotion regulation abilities will be measured using the Emotion Regulation Questionnaire (ERQ), which is composed of 10 items, rated on a 7-point Likert scale, from 0 - strongly disagree to 7 - strongly agree. The scale has two subscales: cognitive reappraisal and expressive suppression emotional regulation strategies. The two subscales had Cronbach's Alphas of .85, respectively .76, similar to those reported in previous studies40.
Changes in emotion regulation | Post-intervention (one week after the intervention)
  Emotion regulation abilities will be measured using the Emotion Regulation Questionnaire (ERQ39), which is composed of 10 items, rated on a 7-point Likert scale, from 0 - strongly disagree to 7 - strongly agree. The scale has two subscales: cognitive reappraisal and expressive suppression emotional regulation strategies. The two subscales had Cronbach's Alphas of .85, respectively .76, similar to those reported in previous studies40.
Levels of emotion regulation | 6 months follow-up
  Emotion regulation abilities will be measured using the Emotion Regulation Questionnaire (ERQ39), which is composed of 10 items, rated on a 7-point Likert scale, from 0 - strongly disagree to 7 - strongly agree. The scale has two subscales: cognitive reappraisal and expressive suppression emotional regulation strategies. The two subscales had Cronbach's Alphas of .85, respectively .76, similar to those reported in previous studies40.
Emotional Distress | Pre-intervention (one week before the intervention)
  Distress and positive emotions: Profile of Affective Distress Plus; PED Opris & Macavei, 2007 is a self-report scale that measure distress. It had 42 items rated on a 5 point Liker scale ranging from "not al all" to "a lot" and grater scores represent grated level of distress.
Changes in emotional distress | Post-intervention (one week after the intervention)
  Distress and positive emotions: Profile of Affective Distress Plus; PED Opris & Macavei, 2007 is a self-report scale that measure distress. It had 42 items rated on a 5 point Liker scale ranging from "not al all" to "a lot" and grater scores represent grated level of distress.
Levels of emotional distress | 6 months follow-up
  Distress and positive emotions: Profile of Affective Distress Plus; PED Opris & Macavei, 2007 is a self-report scale that measure distress. It had 42 items rated on a 5 point Liker scale ranging from "not al all" to "a lot" and grater scores represent grated level of distress.

SECONDARY OUTCOMES:
Mood disorders | baseline, pre-intervention
  The Depression Anxiety Stress Scale (DASS; Parkitny & McAuley, 2010) is a 24 items scale that has three sub scales each measuring a specific problem: depression, anxiety and stress.A higher score at each subscale represents higher levels of depression, anxiety or stress.
Changes in mood disorders | Post-intervention (one week after the intervention)
  The Depression Anxiety Stress Scale (DASS; Parkitny & McAuley, 2010) is a 24 items scale that has three sub scales each measuring a specific problem: depression, anxiety and stress.A higher score at each subscale represents higher levels of depression, anxiety or stress.
Trauma | baseline, pre-intervention
  Childhood Trauma Screener is a scale composed of five items, measuring different traumatic events. It has five items and each item represent a category of trauma. Higher scores represent higher/worse trauma level.

CONTACTS AND LOCATIONS:
Locations (1):
- Babes-Bolyai University, Cluj-Napoca, Romania

IPD SHARING:
Plan to Share IPD: No